CLINICAL TRIAL: NCT02280369
Title: Posture Detection for Automated Abdominal Binder
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 140749
Record Dates: First submitted 2014-09-22; First posted 2014-10-31 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Hypotension, Orthostatic
Keywords: posture detection; healthy subjects
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- automated abdominal binder: automated abdominal binder with waist and thigh accelerometers, and ActivPAL
  Interventions: Device: Automated abdominal binder

INTERVENTIONS:
Device: Automated abdominal binder — Inflatable abdominal binder

SUMMARY:
The automated inflatable abdominal binder is an investigational device for the treatment of orthostatic hypotension (low blood pressure on standing) in autonomic failure patients. The purpose of this study is to evaluate the performance of the binder in detecting body posture during different types of human motion patterns and activities of daily living, and to develop new (and better) ways to detect upright posture. In particular, the investigators want to determine if activities of daily living, normally encountered by patients (lying down, sitting, standing, walking, and climbing up and down steps), interfere with the detection of upright posture used to trigger the device. Studies will be conducted in healthy subjects because the main purpose of this study is to evaluate posture detection rather than treating orthostatic hypotension.

DETAILED DESCRIPTION:
The Primary Objective of this study is to develop and validate the algorithm needed to detect upright posture with a waist 3-axis accelerometer. A Secondary Objective is to determine the performance reliability of posture detection of the thigh and waist accelerometers when exposed to activities of daily living (standing, walking, climbing stairs). We will test the primary and secondary objectives in normal subjects using a single study design. Studies for both objectives will be conducted simultaneously on each subject on a single study day. Normal subjects will wear a device with the waist accelerometer incorporated within the controller box.

Subjects will be instrumented with the abdominal belt and controller box containing the waist accelerometer sensor. The external accelerometer sensor will be fixed with a Velcro around the thigh. In addition, subjects will wear two commercially available accelerometer sensors: 1) the ActivPal on the thigh of the other leg, and 2) an external accelerometer attached to the back of the belt at the level of the waist. The ActivPal can detect the upright posture but cannot distinguish between supine and sitting. The sensor placed on the back will be less affected by belly size in case of obese subjects. Both sensors will be used as a reference and for comparison. We will record all accelerometer signals during different body positions and activities. The activities will include lying down, sitting, getting up and standing still, walking, and climbing up and down steps for about one minute each for a total of 15-20 minutes per group of activities. Participants will perform 3 groups of activities. The order of activities within each group will be randomized. We might also ask you to perform ~3 small jumps to synchronize the sensors at the beginning, middle and the end of each set of activities.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index <30 Kg/m2.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy.
* Any major medical problems or systemic illnesses known to produce orthostatic intolerance.
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing during the screening

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Percentage of times the thigh and waist accelerometer sensors correctly detect upright posture. | during 5-10 minutes performing each activity (lying down, sitting, standing, climbing steps, walking)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States